CLINICAL TRIAL: NCT00796991
Title: A Randomized, Parallel, 3-arm Study to Characterize the Effect of Ipilimumab + Chemotherapy in Patients With Untreated Advanced Melanoma
Brief Title: Drug-Drug Interaction - 3 Arm - Carboplatin/Paclitaxel, Dacarbazine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Medarex (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA184-078
Record Dates: First submitted 2008-11-20; First posted 2008-11-24 (Estimated); Results first posted 2014-01-06 (Estimated); Last update posted 2014-01-06 (Estimated); Status verified 2013-12

CONDITIONS: Advanced Melanoma
Keywords: Untreated Advanced Melanoma
MeSH Terms: interventions — Ipilimumab; Carboplatin; Paclitaxel; BMS 181339; Dacarbazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm A (Active Comparator)
  Interventions: Drug: Ipilimumab; Drug: Carboplatin; Drug: Paclitaxel
- Arm B (Active Comparator)
  Interventions: Drug: Ipilimumab; Drug: Dacarbazine
- Arm C (Active Comparator)
  Interventions: Drug: Ipilimumab

INTERVENTIONS:
Drug: Ipilimumab — Solution, intravenous, 10mg/kg, every 3 weeks in the induction phase, up to 4 doses in the induction phase, 48 weeks
  Other Names: BMS-734016; MDX-010
Drug: Carboplatin — Solution, intravenous, Area Under the Concentration Time Curve=6, every 3 weeks in the induction phase, up to 8 doses in the induction phase, 48 weeks
  Other Names: BMY-26575; PARAPLATIN
  Arms: Arm A
Drug: Paclitaxel — Solution, intravenous, 175 mg/m2, every 3 weeks in the induction phase, up to 8 doses in the induction phase, 48 weeks
  Other Names: TAXOL; BMS-181339
  Arms: Arm A
Drug: Dacarbazine — Solution, intravenous, 850 mg/m2, every 3 weeks in the induction phase, up to 8 doses in the induction phase, 48 weeks
  Arms: Arm B

SUMMARY:
The purpose of this clinical research study is to learn the pharmacokinetics of Ipilimumab when combined with Paclitaxel/Carboplatin or Dacarbazine

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis of advanced malignant melanoma
* Eastern Cooperative Oncology Group (ECOG) performances status 0-1
* Measurable/evaluable disease as per modified World Health Organization (mWHO) criteria

Exclusion Criteria:

* Evidence of active brain metastases
* Prior treatment with anti-cytotoxic lymphocyte antigen 4 (CTLA-4) or anti-CD137 (type of tumor necrosis factor) antibody
* Total Bilirubin greater than (>) 1.5 * upper limit of normal (ULN) and aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 2.5 * upper limit of normal (ULN)
* Prior Autoimmune disease
* Use of immunosuppressing therapies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2009-02; Primary Completion 2009-11 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (4):
- United States (4):
  - The Angeles Clinic & Research Inst., Los Angeles, California
  - H Lee Moffit Cancer Cnt And Res Inst, Tampa, Florida
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Blumenthal Cancer Center, Carolinas Medical Center, Charlotte, North Carolina

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 17 February 2009 study initiated; last patient, last visit (LPLV) 30 October 2012.
Pre-assignment Details: 72 enrolled; 59 randomized and treated with study drug. Reasons for non-randomization: 7 no longer met study criteria; 3 withdrew consent; 1 had target lesion <1 cm; 1 had screening magnetic resonance imaging (MRI) showed brain metastases; 1 had adverse event.
Groups:
- Paclitaxel, Carboplatin, Ipilimumab: Induction Phase: Participant received paclitaxel 175 mg/m^2 intravenously (IV) by a 3-hour infusion and carboplatin IV by a 30-minute infusion) on Day 1 (Week 1, Day 1) and ipilimumab 10 mg/kg IV administered on Day 3 (Week 1, Day 3). Ipilimumab was administered at Weeks 4, 7, and 10, and paclitaxel/carboplatin were administered every 3 weeks (Weeks 4, 7, 10, 13, 16, 19, and 22), with participants receiving the ipilimumab infusion first, followed by the paclitaxel and then carboplatin infusions. A maximum of 8 doses of chemotherapy was permitted. Maintenance Phase: Ipilimumab was administered at a dose of 10 mg/kg every 12 Weeks, beginning at Week 24, until disease progression, study drug-associated toxicity, withdrawal of consent or study closure.
- Dacarbazine, Ipilimumab: Induction Phase: Participant received dacarbazine 850 mg/m^2 IV by a 1-hour infusion on Day 1 (Week 1, Day 1) and ipilimumab at a dose of 10 mg/kg IV administered over 90 minutes on Day 3 (Week 1, Day 3). Ipilimumab was administered at Weeks 4, 7, and 10 and dacarbazine at Weeks 4, 7, 10, 13, 16, 19, and 22), with participants receiving the ipilimumab infusion first, followed by the dacarbazine infusion. A maximum of 8 doses of chemotherapy was permitted. Maintenance Phase: Ipilimumab was administered at a dose of 10 mg/kg every 12 Weeks, beginning at Week 24, until disease progression, study drug-associated toxicity, withdrawal of consent or study closure.
- Ipilimumab: Induction Phase: Participant received ipilimumab at a dose of 10 mg/kg IV administered over 90 minutes every 3 weeks for up to 4 doses (Week 1 Day 1, and Weeks 4, 7, and 10). Maintenance Phase: Ipilimumab was administered at a dose of 10 mg/kg every 12 Weeks, beginning at Week 24, until disease progression, study drug-associated toxicity, withdrawal of consent or study closure.
Period: Overall Study
Arm/Group | Paclitaxel, Carboplatin, Ipilimumab | Dacarbazine, Ipilimumab | Ipilimumab
Started | 20 | 19 | 20
Completed | 5 (Participants continued treatment into maintenance phase.) | 7 (Participants continued treatment into maintenance phase.) | 6 (Participants continued treatment into maintenance phase.)
Not Completed | 15 | 12 | 14
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Death | 2 | 0 | 0
Not completed — Disease Progression | 10 | 9 | 7
Not completed — Study Drug Toxicity | 3 | 3 | 5
Not completed — Withdrawal by Subject | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All randomized and treated participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Paclitaxel, Carboplatin, Ipilimumab | Dacarbazine, Ipilimumab | Ipilimumab | Total
Number analyzed (Participants) | 20 | 19 | 20 | 59
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 15 | 12 | 12 | 39
  >=65 years | 5 | 7 | 8 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (14) | 54 (17) | 60 (11) | 57 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 8 | 21
  Male | 13 | 13 | 12 | 38
Region of Enrollment [Number; unit: participants]
  United States | 20 | 19 | 20 | 59
Eastern Cooperative Oncology Group (ECOG) [Number; unit: participants] — ECOG performance: 0= Fully active, able to carry on all pre-disease performance without restriction;1=Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature; 2=Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours; 3=Capable of only limited self-care, confined to bed or chair more than 50% of waking hours; 4=Completely disabled. Cannot carry on any self-care. Totally confined to bed or Chair; 5=Dead
  participants
    0 | 14 | 17 | 16 | 47
    1 | 6 | 1 | 4 | 11
    2 | 0 | 0 | 0 | 0
    Not Reported | 0 | 1 | 0 | 1
Number of Target Lesions [Number; unit: Participants] — Number of participants with 1, 2, 3, 4, or greater than or equal to (>=) 5 lesions which were targeted for the study.
  Participants
    1 lesion | 4 | 3 | 4 | 11
    2 lesions | 3 | 3 | 0 | 6
    3 lesions | 3 | 4 | 4 | 11
    4 lesions | 0 | 2 | 5 | 7
    >=5 lesions | 10 | 7 | 7 | 24

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetic Parameter Maximum Observed Serum Concentration (Cmax) for Ipilimumab, Paclitaxel, Dacarbazine and the Active Metabolite for Dacarbazine, 5-aminoimidazole-4carboxamide (AIC)- Pharmacokinetic Analysis Population
Description: Cmax=micrograms per milliliter (µg/mL): drug concentration versus time for ipilimumab (Day 43) and paclitaxel, dacarbazine, and AIC (Days 1, 43). Ipilimumab determined from plasma by Enzyme-linked Immunosorbent Assay (ELISA); lower level of quantitation (LLOQ)=0.8 µg/mL; upper limit of quantitation (ULOQ)=25.6 µg/mL; Day 43=0 hour (h) predose, 1.5, 4.0, 24, 72, 168, 336, 504 h post dose; from Day 162 on every 12 weeks (Day 1 and 22= 0 h). Paclitaxel determined using liquid chromatography tandem mass spectrometry (LC/MS/MS) detection; LLOQ=10 nanograms per milliliter (ng/mL); ULOQ=5000 ng/mL; Day 1 and Day 43=0 h predose, 1.5, 3.0, 3.5, 5,5, 9.5, 24, 48 h postdose. Dacarbazine (DTIC) and AIC determined from plasma using liquid chromatography atmospheric pressure ionization (API) tandem mass spectrometry (LC-API/MS/MS) detection; LLOQ for dacarbazine=10.0 ng/mL; ULOQ=5000 ng/mL; AIC LLOQ=0.05 µg/mL; ULOQ=25.0 µg/mL; Day 1: 0 h predose, 1, 1.5, 2.5, 3.5, 5.5, 9.5, 24 h post dose.
Time Frame: Day 1 (0 h) to Day 43
Population: N=participants who received study drug and with adequate Pharmacokinetic (PK) profiles. N is presented for each study drug in each category below. Day 1=paclitaxel/carboplatin or Day 1=dacarbazine; Day 43=ipilimumab+paclitaxel/carboplatin or Day 43=ipilimumab+dacarbazine.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Paclitaxel, Carboplatin, Ipilimumab | Dacarbazine, Ipilimumab | Ipilimumab
Number analyzed (Participants) | 20 | 19 | 12
µg/mL
  Cmax of Ipilimumab N=14, 14, 12 | 234.54 (29) | 246.50 (35) | 251.05 (34)
  Cmax of Paclitaxel (Day 1) N=20, 0, 0 | 3.35 (23) | NA (NA) — Paclitaxel not administered in this arm. | NA (NA) — Paclitaxel not administered in this arm.
  Cmax of Paclitaxel (Day 43) N=14, 0, 0 | 3.19 (26) | NA (NA) — Paclitaxel not administered in this arm. | NA (NA) — Paclitaxel not administered in this arm.
  Cmax of Dacarbazine (Day 1) N=0, 19, 0 | NA (NA) — Dacarbazine not administered in this arm | 18.23 (37) | NA (NA) — Dacarbazine not administered in this arm
  Cmax of Dacarbazine (Day 43) N=0, 16, 0 | NA (NA) — .Dacarbazine not administered in this arm | 18.61 (30) | NA (NA) — Dacarbazine not administered in this arm
  Cmax of AIC (Day 1) N=0, 19, 0 | NA (NA) — Dacarbazine not administered in this arm | 3.57 (36) | NA (NA) — Dacarbazine not administered in this arm
  Cmax of AIC (Day 43) N=0, 17, 0 | NA (NA) — Dacarbazine not administered in this arm | 3.98 (40) | NA (NA) — Dacarbazine not administered in this arm
Statistical Analysis 1: Comparison: Paclitaxel, Carboplatin, Ipilimumab; Estimated effect of ipilimumab on paclitaxel Cmax. Point estimates and 90% confidence intervals (CIs) for means and differences between means on the log scale were exponentiated to obtain estimates for geometric means and ratio of geometric means on the original scale for the paclitaxel/carboplatin/ipilimumab combination (Day 43) relative to paclitaxel/carboplatin alone (Day 1); Test type: Superiority or Other; Mixed Models Analysis; A general linear mixed model was applied to paclitaxel log(Cmax) using study day as a fixed effect; Adjusted geometric mean ratio = 0.963, 90% CI 2-sided [0.794 to 1.168]
Statistical Analysis 2: Comparison: Dacarbazine, Ipilimumab; Estimated effect of ipilimumab on dacarbazine Cmax. Point estimates and 90% confidence intervals (CIs) for means and differences between means on the log scale were exponentiated to obtain estimates for geometric means and ratio of geometric means on the original scale for the dacarbazine, ipilimumab combination (Day 43) relative to dacarbazine alone (Day 1); Test type: Superiority or Other; Mixed Models Analysis; study day was used as a fixed effect; Adjusted geometric mean ratio = 1.027, 90% CI 2-sided [0.848 to 1.243]
Statistical Analysis 3: Comparison: Dacarbazine, Ipilimumab; Estimated effect of ipilimumab on AIC Cmax. Point estimates and 90% confidence intervals (CIs) for means and differences between means on the log scale were exponentiated to obtain estimates for geometric means and ratio of geometric means on the original scale for the dacarbazine, ipilimumab combination (Day 43) relative to dacarbazine alone (Day 1); Test type: Superiority or Other; Mixed Models Analysis; study day was used as a fixed effect; Adjusted geometric mean ratio = 1.058, 90% CI 2-sided [0.974 to 1.150]
Statistical Analysis 4: Comparison: Paclitaxel, Carboplatin, Ipilimumab vs Ipilimumab; Estimated effect of paclitaxel/carboplatin on ipilimumab Cmax: linear model was applied to ipilimumab log(Cmax)) data from Week 7 (Day 43) PK measurements in first and third arms with treatment arm as a fixed effect. Point estimates and 90% CIs for means and differences between means on the log scale were exponentiated to obtain estimates for geometric means and ratio of geometric means on the original scale for the 3 drug combination relative to ipilimumab alone; Test type: Superiority or Other; linear model; treatment arm as a fixed effect; Adjusted geometric mean ratio = 0.934, 90% CI [0.768 to 1.136]
Statistical Analysis 5: Comparison: Dacarbazine, Ipilimumab vs Ipilimumab; Estimated effect of dacarbazine on ipilimumab Cmax: linear model was applied to ipilimumab log(Cmax) data from Week 7 (Day 43) PK measurements in second and third arms with treatment arm as a fixed effect. Point estimates and 90% CIs for means and differences between means on the log scale were exponentiated to obtain estimates for geometric means and ratio of geometric means on the original scale for the dacarbazine, ipilimumab combination relative to ipilimumab alone; Test type: Superiority or Other; linear model; treatment arm as a fixed effect; Adjusted geometric mean ratio = 0.982, 90% CI 2-sided [0.798 to 1.208]

2. Secondary Outcome: Pharmacokinetic Parameter of Time of Maximum Observed Concentration (Tmax) for Ipilimumab, Paclitaxel, Dacarbazine and Active Metabolite AIC - Pharmacokinetic Analysis Population
Description: Tmax reported in hours (h): derived from drug concentration versus time for ipilimumab (Day 43 only) and paclitaxel, dacarbazine, and AIC (Days 1, 43). Ipilimumab determined from plasma ELISA; LLOQ=0.8 µg/mL; ULOQ=25.6 µg/mL; sample times on Day 43=0 hour (h) predose, 1.5, 4.0, 24, 72, 168, 336, 504 h post dose; starting Day 162 every 12 weeks (Day 1 and 22= 0 h). Paclitaxel determined from plasma using LC/MS/MS detection; LLOQ=10 nanograms per milliliter (ng/mL); ULOQ=5000 ng/mL; sample times Day 1 and Day 43=0 h predose, 1.5, 3.0, 3.5, 5,5, 9.5, 24, 48 h postdose. Dacarbazine (DTIC) and AIC determined from plasma using liquid chromatography API tandem mass spectrometry (LC-API/MS/MS) detection; LLOQ for dacarbazine=10.0 ng/mL; ULOQ=5000 ng/mL; AIC LLOQ=0.05 µg/mL; ULOQ=25.0 µg/mL; sample times Day 1: 0 h predose, 1, 1.5, 2.5, 3.5, 5.5, 9.5, 24 h post dose..
Time Frame: Day 1 (0 h) to Day 43
Population: N=participants who received study drug and with adequate PK profiles. N is presented for each study drug in each category below. Day 1=paclitaxel/carboplatin or Day 1=dacarbazine; Day 43=ipilimumab+paclitaxel/carboplatin or Day 43=ipilimumab+dacarbazine.
Measure: Median (Full Range); unit: h
Arm/Group | Paclitaxel, Carboplatin, Ipilimumab | Dacarbazine, Ipilimumab | Ipilimumab
Number analyzed (Participants) | 20 | 19 | 12
h
  Tmax of Ipilimumab N=14, 14, 12 | 1.51 [1.5 to 24.0] | 4.00 [1.5 to 24.6] | 1.56 [1.5 to 4.0]
  Tmax of Paclitaxel (Day 1) N=20, 0, 0 | 3.00 [2.9 to 4.3] | NA [NA to NA] — Paclitaxel not administered in this arm. | NA [NA to NA] — Paclitaxel not administered in this arm.
  Tmax of Paclitaxel (Day 43) N=14, 0, 0 | 3.00 [1.5 to 9.5] | NA [NA to NA] — Paclitaxel not administered in this arm. | NA [NA to NA] — Paclitaxel not administered in this arm.
  Tmax of Dacarbazine (Day 1) N=0, 18, 0 | NA [NA to NA] — Dacarbazine not administered in this arm | 1.00 [1.0 to 2.8] | NA [NA to NA] — Dacarbazine not administered in this arm
  Tmax of Dacarbazine (Day 43) N=0, 15, 0 | NA [NA to NA] — Dacarbazine not administered in this arm | 1.00 [1.0 to 1.1] | NA [NA to NA] — Dacarbazine not administered in this arm
  Tmax of AIC (Day 1) N=0, 19 0 | NA [NA to NA] — Dacarbazine not administered in this arm | 1.00 [1.0 to 2.8] | NA [NA to NA] — Dacarbazine not administered in this arm
  Tmax of AIC (Day 43) N=0, 16, 0 | NA [NA to NA] — Dacarbazine not administered in this arm | 1.00 [1.0 to 2.5] | NA [NA to NA] — Dacarbazine not administered in this arm

3. Secondary Outcome: Pharmacokinetic Parameter of Terminal Elimination Half Life (T-HALF) for Ipilimumab, Paclitaxel, Dacarbazine and Active Metabolite AIC - Pharmacokinetic Analysis Population
Description: T(HALF) reported in hours (h): derived from drug concentration versus time for ipilimumab (Day 43 only) and paclitaxel, dacarbazine, and AIC (Days 1, 43). Ipilimumab determined from plasma ELISA; LLOQ=0.8 µg/mL; ULOQ=25.6 µg/mL; sample times on Day 43=0 hour (h) predose, 1.5, 4.0, 24, 72, 168, 336, 504 h post dose; starting Day 162 every 12 weeks (Day 1 and 22= 0 h). Paclitaxel determined from plasma using LC/MS/MS detection; LLOQ=10 nanograms per milliliter (ng/mL); ULOQ=5000 ng/mL; sample times Day 1 and Day 43=0 h predose, 1.5, 3.0, 3.5, 5,5, 9.5, 24, 48 h postdose. Dacarbazine (DTIC) and AIC determined from plasma using liquid chromatography API tandem mass spectrometry (LC-API/MS/MS) detection; LLOQ for dacarbazine=10.0 ng/mL; ULOQ=5000 ng/mL; AIC LLOQ=0.05 µg/mL; ULOQ=25.0 µg/mL; sample times Day 1: 0 h predose, 1, 1.5, 2.5, 3.5, 5.5, 9.5, 24 h post dose.
Time Frame: Day 1 (0 h) to Day 43
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Paclitaxel, Carboplatin, Ipilimumab | Dacarbazine, Ipilimumab | Ipilimumab
Number analyzed (Participants) | 20 | 19 | 12
h
  T(HALF) of Ipilimumab N=14, 14, 12 | 13.93 (7.54) | 13.39 (4.51) | 15.25 (4.64)
  T(HALF) of Paclitaxel (Day 1) N=20, 0, 0 | 10.26 (1.57) | NA (NA) — Paclitaxel not administered in this arm. | NA (NA) — Paclitaxel not administered in this arm.
  T(HALF) of Paclitaxel (Day 43) N=14, 0, 0 | 10.41 (2.73) | NA (NA) — Paclitaxel not administered in this arm. | NA (NA) — Paclitaxel not administered in this arm.
  T(HALF) of Dacarbazine (Day 1) N=0, 19, 0 | NA (NA) — Dacarbazine not administered in this arm | 2.11 (0.87) | NA (NA) — Dacarbazine not administered in this arm
  T(HALF) of Dacarbazine (Day 43) N=0, 16, 0 | NA (NA) — Dacarbazine not administered in this arm | 2.07 (0.85) | NA (NA) — Dacarbazine not administered in this arm
  T(HALF) of AIC (Day 1) N=0, 18, 0 | NA (NA) — Dacarbazine not administered in this arm | 2.24 (0.96) | NA (NA) — Dacarbazine not administered in this arm
  T(HALF) of AIC (Day 43) N=0, 16, 0 | NA (NA) — Dacarbazine not administered in this arm | 2.21 (0.81) | NA (NA) — Dacarbazine not administered in this arm

4. Secondary Outcome: Pharmacokinetic Parameter of Clearance (CLT) for Ipilimumab, Paclitaxel, Dacarbazine and Active Metabolite AIC - Pharmacokinetic Analysis Population
Description: CLT reported in milliliters/hour (mL/h): derived from drug concentration versus time for ipilimumab (Day 43 only) and paclitaxel, dacarbazine, and AIC (Days 1, 43). Ipilimumab determined from plasma ELISA; LLOQ=0.8 µg/mL; ULOQ=25.6 µg/mL; sample times on Day 43=0 hour (h) predose, 1.5, 4.0, 24, 72, 168, 336, 504 h post dose; starting Day 162 every 12 weeks (Day 1 and 22= 0 h). Paclitaxel determined from plasma using LC/MS/MS detection; LLOQ=10 nanograms per milliliter (ng/mL); ULOQ=5000 ng/mL; sample times Day 1 and Day 43=0 h predose, 1.5, 3.0, 3.5, 5,5, 9.5, 24, 48 h postdose. Dacarbazine (DTIC) and AIC determined from plasma using liquid chromatography API tandem mass spectrometry (LC-API/MS/MS) detection; LLOQ for dacarbazine=10.0 ng/mL; ULOQ=5000 ng/mL; AIC LLOQ=0.05 µg/mL; ULOQ=25.0 µg/mL; sample times Day 1: 0 h predose, 1, 1.5, 2.5, 3.5, 5.5, 9.5, 24 h post dose..
Time Frame: Day 1 (0 h) to Day 43
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/h
Arm/Group | Paclitaxel, Carboplatin, Ipilimumab | Dacarbazine, Ipilimumab | Ipilimumab
Number analyzed (Participants) | 20 | 19 | 12
mL/h
  CLT of Ipilimumab N=14, 14, 12 | 11.63 (50) | 11.17 (34) | 10.23 (44)
  CLT of Paclitaxel (Day 1) N=20, 0, 0 | 27.87 (28) | NA (NA) — Paclitaxel not administered in this arm. | NA (NA) — Paclitaxel not administered in this arm.
  CLT of Paclitaxel (Day 43) N=14, 0, 0 | 25.44 (26) | NA (NA) — Paclitaxel not administered in this arm. | NA (NA) — Paclitaxel not administered in this arm.
  CLT of Dacarbazine (Day 1) N=0, 19, 0 | NA (NA) — Dacarbazine not administered in this arm | 34.33 (52) | NA (NA) — Dacarbazine not administered in this arm
  CLT of Dacarbazine (Day 43) N=0, 16, 0 | NA (NA) — Dacarbazine not administered in this arm | 37.09 (49) | NA (NA) — Dacarbazine not administered in this arm
  CLT of AIC (Day 1) N=0, 19, 0 | NA (NA) — Dacarbazine not administered in this arm | 91.67 (28) | NA (NA) — Dacarbazine not administered in this arm
  CLT of AIC (Day 43) N=0, 17, 0 | NA (NA) — Dacarbazine not administered in this arm | 88.75 (37) | NA (NA) — Dacarbazine not administered in this arm

5. Primary Outcome: Area Under the Concentration Time Curve (AUC) From Time Zero to 21 Days [AUC(0-21d)] for Ipilimumab and AUC Time Zero Extrapolated to Infinity [AUC(INF)] for Paclitaxel, Dacarbazine and the Active Metabolite AIC - Pharmacokinetic Analysis Population
Description: AUC=micrograms*hour(h) per mL (µg*h/mL): derived from drug concentration versus time for ipilimumab (Day 43 only) and paclitaxel, dacarbazine, and AIC (Days 1, 43). Ipilimumab determined from plasma ELISA; LLOQ=0.8 µg/mL; ULOQ=25.6 µg/mL; sample times on Day 43=0 hour (h) predose, 1.5, 4.0, 24, 72, 168, 336, 504 h post dose; starting Day 162 every 12 weeks (Day 1 and 22= 0 h). Paclitaxel determined from plasma using LC/MS/MS detection; LLOQ=10 nanograms per milliliter (ng/mL); ULOQ=5000 ng/mL; sample times Day 1 and Day 43=0 h predose, 1.5, 3.0, 3.5, 5,5, 9.5, 24, 48 h postdose. Dacarbazine (DTIC) and AIC determined from plasma using liquid chromatography API tandem mass spectrometry (LC-API/MS/MS) detection; LLOQ for dacarbazine=10.0 ng/mL; ULOQ=5000 ng/mL; AIC LLOQ=0.05 µg/mL; ULOQ=25.0 µg/mL; sample times Day 1: 0 h predose, 1, 1.5, 2.5, 3.5, 5.5, 9.5, 24 h post dose.
Time Frame: Day 1 (0 h) to Day 43
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg*h/mL
Arm/Group | Paclitaxel, Carboplatin, Ipilimumab | Dacarbazine, Ipilimumab | Ipilimumab
Number analyzed (Participants) | 20 | 19 | 12
µg*h/mL
  AUC(0-21d) of Ipilimumab N=14, 14, 12 | 46925.36 (36) | 49569.06 (25) | 54039.79 (28)
  AUC(INF) of Paclitaxel (Day 1) N=20, 0, 0 | 12.37 (24) | NA (NA) — Paclitaxel not administered in this arm. | NA (NA) — Paclitaxel not administered in this arm.
  AUC(INF) of Paclitaxel (Day 43) N=14, 0, 0 | 13.41 (24) | NA (NA) — Paclitaxel not administered in this arm. | NA (NA) — Paclitaxel not administered in this arm.
  AUC(INF) of Dacarbazine (Day 1) N=0, 19, 0 | NA (NA) — Dacarbazine not administered in this arm. | 47.36 (68) | NA (NA) — Dacarbazine not administered in this arm.
  AUC(INF) of Dacarbazine (Day 43) N=0, 16, 0 | NA (NA) — Dacarbazine not administered in this arm. | 41.13 (55) | NA (NA) — Dacarbazine not administered in this arm.
  AUC(INF) of AIC (Day 1) N=0, 18, 0 | NA (NA) — Dacarbazine not administered in this arm. | 17.68 (26) | NA (NA) — Dacarbazine not administered in this arm.
  AUC(INF) of AIC (Day 43) N=0, 16, 0 | NA (NA) — Dacarbazine not administered in this arm. | 17.38 (36) | NA (NA) — Dacarbazine not administered in this arm.
Statistical Analysis 1: Comparison: Paclitaxel, Carboplatin, Ipilimumab; Estimated effect of ipilimumab on paclitaxel AUC(INF). Point estimates and 90% confidence intervals (CIs) for means and differences between means on the log scale were exponentiated to obtain estimates for geometric means and ratio of geometric means on the original scale for the paclitaxel/carboplatin/ipilimumab combination (Day 43) relative to paclitaxel/carboplatin alone (Day 1); Test type: Superiority or Other; Mixed Models Analysis; A general linear mixed model was applied to paclitaxel log[AUC(INF)] using study day as a fixed effect; Geometric mean ratio = 1.068, 90% CI 2-sided [0.954 to 1.196]
Statistical Analysis 2: Comparison: Dacarbazine, Ipilimumab; Estimated effect of ipilimumab on dacarbazine AUC(INF). Point estimates and 90% confidence intervals (CIs) for means and differences between means on the log scale were exponentiated to obtain estimates for geometric means and ratio of geometric means on the original scale for the dacarbazine, ipilimumab combination (Day 43) relative to dacarbazine alone (Day 1); Test type: Superiority or Other; Mixed Models Analysis; A general linear mixed model was applied to dacarbazine log[AUC(INF)] using study day as a fixed effect; Adjusted geometric mean ratio = 0.912, 90% CI 2-sided [0.757 to 1.099]
Statistical Analysis 3: Comparison: Dacarbazine, Ipilimumab; Estimated effect of ipilimumab on AUC(INF) for AIC. Point estimates and 90% confidence intervals (CIs) for means and differences between means on the log scale were exponentiated to obtain estimates for geometric means and ratio of geometric means on the original scale for the dacarbazine, ipilimumab combination (Day 43) relative to dacarbazine alone (Day 1); Test type: Superiority or Other; Mixed Models Analysis; A general linear mixed model was applied to active metabolite AIC log[AUC(INF)] using study day as a fixed effect; Adjusted geometric mean ratio = 0.970, 90% CI 2-sided [0.891 to 1.056]
Statistical Analysis 4: Comparison: Paclitaxel, Carboplatin, Ipilimumab vs Ipilimumab; Estimated effect of paclitaxel/carboplatin on ipilimumab AUC: linear model was applied to ipilimumab log(AUC(0-21d)) data from Week 7 (Day 43) PK measurements in first and third arms with treatment arm as a fixed effect. Point estimates and 90% CIs for means and differences between means on the log scale were exponentiated to obtain estimates for geometric means and ratio of geometric means on the original scale for the 3 drug combination relative to ipilimumab alone; Test type: Superiority or Other; linear model; treatment arm as fixed effect; Adjusted geometric mean ratio = 0.934, 90% CI 2-sided [0.768 to 1.136]
Statistical Analysis 5: Comparison: Dacarbazine, Ipilimumab vs Ipilimumab; Estimated effect of dacarbazine on ipilimumab AUC: linear model was applied to ipilimumab log(AUC(0-21d)) data from Week 7 (Day 43) PK measurements in second and third arms with treatment arm as a fixed effect. Point estimates and 90% CIs for means and differences between means on the log scale were exponentiated to obtain estimates for geometric means and ratio of geometric means on the original scale for the dacarbazine, ipilimumab combination relative to ipilimumab alone; Test type: Superiority or Other; linear model; treatment arm as a fixed effect; Adjusted geometric mean ratio = 0.982, 90% CI 2-sided [0.7981 to 1.208]

6. Secondary Outcome: Pharmacokinetic Parameter Volume of Distribution at Steady State (Vss) for Ipilimumab, Paclitaxel, Dacarbazine and Active Metabolite AIC - Pharmacokinetic Analysis Population
Description: Vss reported in liters(L): derived from drug concentration versus time for ipilimumab (Day 43 only) and paclitaxel, dacarbazine, and AIC (Days 1, 43). Ipilimumab determined from plasma ELISA; LLOQ=0.8 µg/mL; ULOQ=25.6 µg/mL; sample times on Day 43=0 hour (h) predose, 1.5, 4.0, 24, 72, 168, 336, 504 h post dose; starting Day 162 every 12 weeks (Day 1 and 22= 0 h). Paclitaxel determined from plasma using LC/MS/MS detection; LLOQ=10 nanograms per milliliter (ng/mL); ULOQ=5000 ng/mL; sample times Day 1 and Day 43=0 h predose, 1.5, 3.0, 3.5, 5,5, 9.5, 24, 48 h postdose. Dacarbazine (DTIC) and AIC determined from plasma using liquid chromatography API tandem mass spectrometry (LC-API/MS/MS) detection; LLOQ for dacarbazine=10.0 ng/mL; ULOQ=5000 ng/mL; AIC LLOQ=0.05 µg/mL; ULOQ=25.0 µg/mL; sample times Day 1: 0 h predose, 1, 1.5, 2.5, 3.5, 5.5, 9.5, 24 h post dose.
Time Frame: Day 1 (0 h) to Day 43
Population: N=participants who received study drug and with adequate PK profiles. N is presented for each study drug in each category below. Day 43=ipilimumab+paclitaxel/carboplatin or Day 43=ipilimumab+dacarbazine.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | Paclitaxel, Carboplatin, Ipilimumab | Dacarbazine, Ipilimumab | Ipilimumab
Number analyzed (Participants) | 20 | 19 | 12
L
  Vss of Ipilimumab N=14, 14, 12 | 5.10 (25) | 4.88 (21) | 5.05 (29)
  Vss of Paclitaxel (Day 43) N=14, 0, 0 | 205.63 (31) | NA (NA) — Paclitaxel not administered in this arm. | NA (NA) — Paclitaxel not administered in this arm.
  Vss of Dacarbazine (Day 43) N=0, 16, 0 | NA (NA) — Dacarbazine not administered in this arm. | 107.90 (31) | NA (NA) — Dacarbazine not administered in this arm.
  Vss of AIC (Day 1) N=0, 17, 0 | NA (NA) — Dacarbazine not administered in this arm. | 342.64 (47) | NA (NA) — Dacarbazine not administered in this arm.

7. Secondary Outcome: Number of Participants in Best Overall Response Categories Based on Modified World Health Organization (mWHO) Criteria - All Treated Participants
Description: Assessments for antitumor activity by physical exam and routine anatomic imaging were at Week 12 and confirmatory imaging at Weeks 16, 20, and 24. Participants with resected index or new lesions were considered progressed in their disease. Complete Response (CR): Complete disappearance of all index lesions; Partial Response (PR): Decrease, relative to baseline, of 50% or greater in the sum of the products of the two largest perpendicular diameters of all index lesions, in the absence of Complete Response; Stable Disease (SD): Does not meet criteria for complete or partial response, in the absence of progressive disease. Participants with PR or CR that was not confirmed after at least 4 weeks are scored as SD unless they have new primary lesions; Progressive Disease: At least 25% increase in the sum of products of all index lesions and/or the appearance of any new lesion(s). Unknown=the participants overall response was not known.
Time Frame: Day 1 to Week 48
Population: Treated participants received at least one dose of a study drug.
Measure: Number; unit: participants
Arm/Group | Paclitaxel, Carboplatin, Ipilimumab | Dacarbazine, Ipilimumab | Ipilimumab
Number analyzed (Participants) | 20 | 19 | 20
participants
  Complete Response | 1 | 1 | 0
  Partial Response | 1 | 4 | 5
  Stable Disease | 6 | 5 | 4
  Progressive Disease | 9 | 8 | 8
  Unknown | 3 | 1 | 3

8. Secondary Outcome: Number of Participants in Best Overall Response Categories Based on Immune Related (ir) Response Criteria (RC) - All Treated Participants
Description: Assessments: Weeks 12, 16, 20, and 24. Participants with resected index or new lesions considered progressed in their disease. The immune-related (ir) response criteria (irRC) represents further modifications of mWHO criteria reflecting clinical experience with ipilimumab in which objective and durable responses (as per mWHO) were observed in participants following progression and without intervening alternative anti-cancer therapy. Immune-related (ir)Complete Response (irCR): Complete disappearance of all index lesions; ir Partial Response (irPR): Decrease, relative to baseline, of 50% or greater in sum of products of the two largest perpendicular diameters of all index and all new measurable lesions, in the absence of irCR; ir Stable Disease (irSD): Does not meet criteria for irCR or irPR, in the absence of progressive disease (PD); ir PD: At least 25% increase in Tumor Burden compared to sum of product diameters (SPD) at nadir. ir Unknown=participants overall response not known.
Time Frame: Day 1 to Week 48
Population: Treated participants received at least one dose of a study drug.
Measure: Number; unit: participants
Arm/Group | Paclitaxel, Carboplatin, Ipilimumab | Dacarbazine, Ipilimumab | Ipilimumab
Number analyzed (Participants) | 20 | 19 | 20
participants
  ir Complete Response | 1 | 1 | 0
  ir Partial Response | 4 | 5 | 5
  ir Stable Disease | 5 | 5 | 6
  ir Progressive Disease | 7 | 7 | 6
  ir Unknown | 3 | 1 | 3

9. Secondary Outcome: Number of Participants With Objective Response to Treatment and Disease Control Using mWHO Criteria - All Randomized Participants
Description: Number of participants with an objective response to treatment excluded participants with a best overall response (BOR) of Stable Disease (SD). Disease control is non-progression of disease while on treatment. A participant was considered to have achieved disease control if he/she had a BOR of CR, PR, or SD in the absence of resected index lesions or new lesions while the participant was considered to have an objective response to treatment in he/she had a BOR of CR or PR in the absence of resected index lesions or new lesions.
Time Frame: Day 1 to Week 48
Population: Randomized Population includes all participants randomized to a treatment arm
Measure: Number; unit: participants
Arm/Group | Paclitaxel, Carboplatin, Ipilimumab | Dacarbazine, Ipilimumab | Ipilimumab
Number analyzed (Participants) | 20 | 19 | 20
participants
  Participants with Objective Response | 2 | 5 | 5
  Participants with Disease Control | 8 | 10 | 9

10. Secondary Outcome: Number of Participants With Adverse Events, Serious Adverse Events, Deaths, and Discontinuation Due to Adverse Events From Day 1 to Week 48 - All Treated Population
Description: Adverse events (AEs) and Serious AEs (SAEs) were graded using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse events version 3.0. Week 48 database lock was 27 July 2010.
Time Frame: Day 1 to Week 48
Population: Treated participants received at least one dose of a study drug.
Measure: Number; unit: participants
Arm/Group | Paclitaxel, Carboplatin, Ipilimumab | Dacarbazine, Ipilimumab | Ipilimumab
Number analyzed (Participants) | 20 | 19 | 20
participants
  Participants with AEs | 20 | 19 | 20
  Participants with SAEs | 9 | 8 | 9
  Participants with SAEs Treatment-Related | 4 | 6 | 5
  Deaths | 12 | 5 | 7
  Deaths Treatment-Related | 0 | 0 | 0
  Participants discontinued due to AE(s) | 6 | 7 | 5

11. Secondary Outcome: Mean Absolute Lymphocyte Count (ALC) at Each Nominal Ipilimumab Induction Dose and at End of the Induction Period - Pharmacodynamic Population
Description: Absolute lymphocyte counts were obtained from routine hematology panels from 28 days prior to the first treatment with any study medication through the end of the Induction-Dosing Period and were reported as number*10^3 cells per micro liter (x10^3 c/µL).
Time Frame: Day to Week 12
Population: Pharmacodynamic Population: All treated participants with one unambiguous date of first dose; and at least 1 ALC evaluation during the induction-dosing period. For each of these participants, all ALC evaluations from 28 days prior to first dose of any study medication to the end of the induction dosing are included.
  period.
Measure: Mean (95% Confidence Interval); unit: 10^3 cells/µL
Arm/Group | Paclitaxel, Carboplatin, Ipilimumab | Dacarbazine, Ipilimumab | Ipilimumab
Number analyzed (Participants) | 29 | 19 | 20
10^3 cells/µL
  Nominal Ipilimumab Induction Dose Number 1 | 1.19 [0.79 to 1.59] | 1.41 [1.00 to 1.82] | 1.28 [0.91 to 1.64]
  Nominal Ipilimumab Induction Dose Number 2 | 1.62 [1.27 to 1.98] | 2.05 [1.69 to 2.42] | 1.56 [1.18 to 1.93]
  Nominal Ipilimumab Induction Dose Number 3 | 1.43 [1.06 to 1.80] | 1.96 [1.59 to 2.33] | 1.99 [1.59 to 2.39]
  Nominal Ipilimumab Induction Dose Number 4 | 1.42 [1.03 to 1.80] | 1.87 [1.49 to 2.25] | 1.80 [1.39 to 2.22]
  End of Ipilimumab Induction dosing Period | 1.67 [1.23 to 2.10] | 2.07 [1.63 to 2.51] | 1.73 [1.20 to 2.25]
Statistical Analysis 1: Comparison: Paclitaxel, Carboplatin, Ipilimumab vs Dacarbazine, Ipilimumab vs Ipilimumab; null hypothesis of no mean ALC changes over time in any treatment group. Conditional F-tests were used to test for mean ALC changes over time in each treatment arm and the difference between treatment arms in the pattern of change in ALC over time; Test type: Superiority or Other; p = 0.027, conditional F test — p-value was not corrected for multiple testing. F-statistic = 1.86; 15 degrees freedom (DF) in numerator and 335 DF in denominator
Statistical Analysis 2: Comparison: Paclitaxel, Carboplatin, Ipilimumab vs Dacarbazine, Ipilimumab vs Ipilimumab; null hypothesis that the pattern of mean ALC values over time is the same in all treatment groups. Test of overall time-by-treatment interaction used an omnibus conditional F-test; Test type: Superiority or Other; p = 0.5, Omnibus conditional F-test — P-values were not corrected for multiple testing. F Statistic =0.94; 10 Degrees Freedom (DF) in numerator and 335 DF in denominator
Statistical Analysis 3: Comparison: Paclitaxel, Carboplatin, Ipilimumab vs Ipilimumab; null hypothesis that the pattern of mean ALC values over time is the same in the given pair of treatment groups; Test type: Superiority or Other; p = 0.37, conditional F-test — P-values were not corrected for multiple testing. F Statistic =1.08; 5 Degrees Freedom (DF) in numerator and 335 DF in denominator
Statistical Analysis 4: Comparison: Paclitaxel, Carboplatin, Ipilimumab vs Dacarbazine, Ipilimumab; null hypothesis that the pattern of mean ALC values over time is the same in the given pair of treatment groups; Test type: Superiority or Other; p = 0.85, conditional F-test — P-values were not corrected for multiple testing. F Statistic =0.39; 5 Degrees Freedom (DF) in numerator and 335 DF in denominator
Statistical Analysis 5: Comparison: Dacarbazine, Ipilimumab vs Ipilimumab; null hypothesis that the pattern of mean ALC values over time is the same in the given pair of treatment groups; Test type: Superiority or Other; p = 0.22, conditional F-test — P-values were not corrected for multiple testing. F Statistic = 1.41; 5 Degrees Freedom (DF) in numerator and 335 DF in denominator

12. Secondary Outcome: Mean Change From Baseline at Weeks 16 and 48 in Diastolic and Systolic Blood Pressure - All Treated Population
Description: Blood pressure was obtained while the participant was sitting down and was measured in millimeters of mercury (mmHg). During the induction phase blood pressure was collected 30 minutes prior to dosing and every 30 minutes for the duration of the ipilimumab infusion. Orthostatic blood pressure was to be measured when clinically indicated (for example, participant was experiencing lightheadedness, dizziness, syncope). Blood pressures were recorded at Weeks 1, 4, 7, 10,13, 16, 19, and 22 during the Induction Phase, and at Weeks 24, 36, and 48 during the Maintenance Phase.
Time Frame: Day 1 to Week 48
Population: Treated participants received at least one dose of a study drug. N=number of treated participants who also had blood pressure value available for analysis.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Paclitaxel, Carboplatin, Ipilimumab | Dacarbazine, Ipilimumab | Ipilimumab
Number analyzed (Participants) | 1 | 6 | 9
mmHg
  Diastolic Blood Pressure at Week 16 (N=1, 6, 9) | 10.0 (NA) — N=1 so since only 1 participant was analyzed there can be no standard deviation. | 6.6 (11.3) | 4.9 (13.3)
  Diastolic Blood Pressure at Week 48 (N=1, 4, 4) | 2.0 (NA) — N=1 so since only 1 participant was analyzed there can be no standard deviation. | 7.0 (11.3) | 8.5 (8.2)
  Systolic Blood Pressure at Week 16 (N=1, 6, 9) | 22.0 (NA) — N=1 so since only 1 participant was analyzed there can be no standard deviation. | 2.7 (12.2) | 9.7 (14.1)
  Systolic Blood Pressure at Week 48 (N=1, 4, 4) | 5.0 (NA) — N=1 so since only 1 participant was analyzed there can be no standard deviation. | 1.0 (17.1) | 12.0 (8.6)

13. Secondary Outcome: Mean Change From Baseline in Pulse Rate at Weeks 16 and 48 - All Treated Population
Description: Pulse rate was obtained while the participant was sitting down and measured in beats per minute (bpm). During the induction phase pulse rate was collected 30 minutes prior to dosing and every 30 minutes for the duration of the ipilimumab infusion. Pulse rate was recorded at Weeks 1, 4, 7, 10, 13, 16, 19, and 22 during the Induction Phase, and at Weeks 24, 36, and 48 during the Maintenance Phase.
Time Frame: Day 1 to Week 48
Population: Treated participants received at least one dose of a study drug. N=number of treated participants who also had a Pulse rate value available for analysis.
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Paclitaxel, Carboplatin, Ipilimumab | Dacarbazine, Ipilimumab | Ipilimumab
Number analyzed (Participants) | 1 | 6 | 9
bpm
  Pulse Rate at Week 16 (N=1, 6, 9) | 24.0 (NA) — N=1 so since only 1 participant was analyzed there can be no standard deviation. | 0.3 (13.9) | -0.7 (15.9)
  Pulse Rate at Week 48 (N=1, 4, 4) | -3.0 (NA) — N=1 so since only 1 participant was analyzed there can be no standard deviation. | -9.5 (13.6) | 7.5 (10.3)

14. Secondary Outcome: Mean Change From Baseline in Respiration Rate at Weeks 16 and 48 - All Treated Population
Description: Respiration rate was obtained while the participant was sitting down and measured in breaths per minute (bpm). During the induction phase respiration rate was collected 30 minutes prior to dosing and every 30 minutes for the duration of the ipilimumab infusion. Respiration rate was recorded at Weeks 1, 4, 7, 10, 13, 16, 19, and 22 during the Induction Phase, and at Weeks 24, 36, and 48 during the Maintenance Phase.
Time Frame: Day 1 to Week 48
Population: Treated participants received at least one dose of a study drug. N=number of treated participants who also had a Respiration rate value available for analysis.
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Paclitaxel, Carboplatin, Ipilimumab | Dacarbazine, Ipilimumab | Ipilimumab
Number analyzed (Participants) | 1 | 5 | 6
bpm
  Respiration Rate at Week 16 (N=1, 5, 6) | 0 (NA) — N=1 so since only 1 participant was analyzed there can be no standard deviation | 1.4 (2.4) | -0.8 (2.2)
  Respiration Rate at Week 48 (N=1, 3, 3) | -2.0 (NA) — N=1 so since only 1 participant was analyzed there can be no standard deviation | -2.7 (1.2) | -1.3 (1.2)

15. Secondary Outcome: Mean Baseline Change in Body Temperature at Weeks 16 and 48 - All Treated Population
Description: Temperature was obtained while the participant was sitting down and was measured in degrees Fahrenheit (F). During the induction phase this vital sign was collected 30 minutes prior to dosing and every 30 minutes for the duration of the ipilimumab infusion. Temperature was recorded at Weeks 1, 4, 7, 10, 13, 16, 19, and 22 during the Induction Phase, and at Weeks 24, 36, and 48 during the Maintenance Phase.
Time Frame: Day 1 to Week 48
Population: Treated participants received at least one dose of a study drug. N=number of treated participants who also had a temperature value available for analysis.
Measure: Mean (Standard Deviation); unit: degrees F
Arm/Group | Paclitaxel, Carboplatin, Ipilimumab | Dacarbazine, Ipilimumab | Ipilimumab
Number analyzed (Participants) | 20 | 19 | 20
degrees F
  Temperature at Week 16 (N=1, 6, 9) | -0.5 (NA) — N=1 so since only 1 participant was analyzed there can be no standard deviation. | -0.1 (0.8) | 0.2 (0.9)
  Temperature at Week 48 (N=1, 4, 4) | 0.4 (NA) — N=1 so since only 1 participant was analyzed there can be no standard deviation. | 0.0 (0.7) | -0.2 (0.7)

16. Secondary Outcome: Number of Participants on Treatment With Toxicity Changes From Baseline by Worst Common Terminology Criteria (CTC) Grade for Hemoglobin - All Treated Population
Description: Hemoglobin was measured in grams per deciliter (g/dL). National Cancer Institute Common Terminology Criteria (CTC) v3.0 was used to determine Grade. GRADE (1): 10.0 - less than (<) lower limit of normal (LLN); GRADE (2): 8.0 - < 10.0; GRADE (3): 6.5 - < 8.0; GRADE (4): < 6.5
Time Frame: Day 1 to Week 48
Measure: Number; unit: participants
Arm/Group | Paclitaxel, Carboplatin, Ipilimumab | Dacarbazine, Ipilimumab | Ipilimumab
Number analyzed (Participants) | 20 | 19 | 20
participants
  Hemoglobin Grade 0 | 3 | 4 | 5
  Hemoglobin Grade 1 | 9 | 13 | 10
  Hemoglobin Grade 2 | 8 | 1 | 4
  Hemoglobin Grade 3 | 0 | 1 | 0
  Hemoglobin Not Reported | 0 | 0 | 1

17. Secondary Outcome: Number of Participants on Treatment With Toxicity Changes From Baseline by Worst Common Terminology Criteria (CTC) Grade for Leukocytes - All Treated Population
Description: Leukocytes are measured as *10^3 cells per microliter (c/µL). National Cancer Institute Common Terminology Criteria (CTC) version (v) 3.0 was used to determine Grade. GRADE (1): 3.0 - < LLN; GRADE (2): 2.0 - < 3.0; GRADE (3): 1.0 - < 2.0; GRADE (4): < 1.0.
Time Frame: Day 1 to Week 48
Population: Treated participants received at least one dose of a study drug.
Measure: Number; unit: participants
Arm/Group | Paclitaxel, Carboplatin, Ipilimumab | Dacarbazine, Ipilimumab | Ipilimumab
Number analyzed (Participants) | 20 | 19 | 20
participants
  Leukocytes Grade 0 | 8 | 13 | 17
  Leukocytes Grade 1 | 4 | 4 | 1
  Leukocytes Grade 2 | 2 | 2 | 1
  Leukocytes Grade 3 | 5 | 0 | 0
  Leukocytes Grade 4 | 1 | 0 | 0
  Leukocytes Not Reported | 0 | 0 | 1

18. Secondary Outcome: Number of Participants on Treatment With Toxicity Changes From Baseline by Worst Common Terminology Criteria (CTC) Grade for Lymphocytes - All Treated Population
Description: Lymphocytes (absolute) were measured as *10^3 cells per microliter (c/µL). National Cancer Institute Common Terminology Criteria (CTC) version (v) 3.0 was used to determine Grade. GRADE (1): 0.8 - < 1.5; GRADE (2): 0.5 - < 0.8; GRADE (3): 0.2 - < 0.5; GRADE (4): < 0.2
Time Frame: Day 1 to Week 48
Population: Treated participants received at least one dose of a study drug.
Measure: Number; unit: participants
Arm/Group | Paclitaxel, Carboplatin, Ipilimumab | Dacarbazine, Ipilimumab | Ipilimumab
Number analyzed (Participants) | 20 | 19 | 20
participants
  Lymphocytes Grade 0 | 4 | 5 | 6
  Lymphocytes Grade 1 | 12 | 13 | 11
  Lymphocytes Grade 2 | 3 | 1 | 3
  Lymphocytes Grade 3 | 1 | 0 | 0

19. Secondary Outcome: Number of Participants on Treatment With Toxicity Changes From Baseline by Worst CTC Grade for Neutrophils - All Treated Population
Description: Neutrophils (absolute) are measured as *10^3 cells per microliter (c/µL). National Cancer Institute Common Terminology Criteria (CTC) v3.0 was used to determine Grade. GRADE (1): 1.5 - < 2.0; GRADE (2): 1.0 - < 1.5; GRADE (3): 0.5 - < 1.0; GRADE (4): < 0.5
Time Frame: Day 1 to Week 48
Population: Treated participants received at least one dose of a study drug.
Measure: Number; unit: participants
Arm/Group | Paclitaxel, Carboplatin, Ipilimumab | Dacarbazine, Ipilimumab | Ipilimumab
Number analyzed (Participants) | 20 | 19 | 20
participants
  Neutrophils Grade 0 | 20 | 18 | 19
  Neutrophils Grade 1 | 0 | 0 | 1
  Neutrophils Grade 3 | 0 | 1 | 0

20. Secondary Outcome: Number of Participants on Treatment With Toxicity Changes From Baseline by Worst CTC Grade for Neutrophils Plus Bands - All Treated Population
Description: Neutrophils plus bands (absolute) were measured as *10^3 cells per microliter (c/µL). National Cancer Institute Common Terminology Criteria (CTC) v3.0 was used to determine Grade. GRADE (1): 1.5 - < 2.0; GRADE (2): 1.0 - < 1.5; GRADE (3): 0.5 - < 1.0; GRADE (4): < 0.5.
Time Frame: Day 1 to Week 48
Measure: Number; unit: participants
Arm/Group | Paclitaxel, Carboplatin, Ipilimumab | Dacarbazine, Ipilimumab | Ipilimumab
Number analyzed (Participants) | 20 | 19 | 20
participants
  Neutrophils Plus Bands Grade 0 | 20 | 18 | 19
  Neutrophils Plus Bands Grade 1 | 0 | 0 | 1
  Neutrophils Plus Bands Grade 3 | 0 | 1 | 0

21. Secondary Outcome: Number of Participants on Treatment With Toxicity Changes From Baseline by Worst CTC Grade for Platelet Count - All Treated Population
Description: Platelets were measured as *10^9 cells per liter (c/L). National Cancer Institute Common Terminology Criteria (CTC) v3.0 was used to determine Grade. GRADE (1): 75.0 - < LLN; GRADE (2): 50.0 - < 75.0; GRADE (3): 25.0 - < 50.0; GRADE (4): < 25.0.
Time Frame: Day 1 to Week 48
Population: Treated participants received at least one dose of a study drug.
Measure: Number; unit: participants
Arm/Group | Paclitaxel, Carboplatin, Ipilimumab | Dacarbazine, Ipilimumab | Ipilimumab
Number analyzed (Participants) | 20 | 19 | 20
participants
  Platelet Count Grade 0 | 20 | 19 | 18
  Platelet Count Grade 1 | 0 | 0 | 2

22. Secondary Outcome: Number of Participants on Treatment With Toxicity Changes From Baseline by Worst CTC Grade for Alanine Aminotransferase (ALT) - All Treated Population
Description: ALT was measured as Units per Liter (U/L). National Cancer Institute Common Terminology Criteria (CTC) v3.0 was used to determine Grade. GRADE (1): > 1.0 - 2.5 * upper limits of normal (ULN); GRADE (2): > 2.5 - 5.0 * ULN; GRADE (3): > 5.0 - 20.0 * ULN; GRADE (4): > 20.0 * ULN.
Time Frame: Day 1 to Week 48
Population: Treated participants received at least one dose of a study drug.
Measure: Number; unit: participants
Arm/Group | Paclitaxel, Carboplatin, Ipilimumab | Dacarbazine, Ipilimumab | Ipilimumab
Number analyzed (Participants) | 20 | 19 | 20
participants
  ALT Grade 0 | 18 | 18 | 16
  ALT Grade 1 | 2 | 1 | 3
  ALT Grade 2 | 0 | 0 | 1

23. Secondary Outcome: Number of Participants on Treatment With Toxicity Changes From Baseline by Worst CTC Grade for Aspartate Aminotransferase (AST) - All Treated Population
Description: AST was measured as Units per Liter (U/L). National Cancer Institute Common Terminology Criteria (CTC) v3.0 was used to determine Grade. GRADE (1): > 1.0 - 2.5 * upper limits of normal (ULN); GRADE (2): > 2.5 - 5.0 * ULN; GRADE (3): > 5.0 - 20.0 * ULN; GRADE (4): > 20.0 * ULN.
Time Frame: Day 1 to Week 48
Measure: Number; unit: participants
Arm/Group | Paclitaxel, Carboplatin, Ipilimumab | Dacarbazine, Ipilimumab | Ipilimumab
Number analyzed (Participants) | 20 | 19 | 20
participants
  AST Grade 0 | 18 | 18 | 15
  AST Grade 1 | 2 | 1 | 4
  AST Grade 2 | 0 | 0 | 1

24. Secondary Outcome: Number of Participants on Treatment With Toxicity Changes From Baseline by Worst CTC Grade for Albumin - All Treated Population
Description: Albumin was measured in grams per deciliter (g/dL). National Cancer Institute Common Terminology Criteria (CTC) v3.0 was used to determine Grade. GRADE (1): < LLN - 3.0; GRADE (2): < 3.0 - 2.0; GRADE (3): < 2.0 g/dL.
Time Frame: Day 1 to Week 48
Measure: Number; unit: participants
Arm/Group | Paclitaxel, Carboplatin, Ipilimumab | Dacarbazine, Ipilimumab | Ipilimumab
Number analyzed (Participants) | 20 | 19 | 20
participants
  Albumin Grade 0 | 17 | 14 | 14
  Albumin Grade 1 | 3 | 5 | 6

25. Secondary Outcome: Number of Participants on Treatment With Toxicity Changes From Baseline by Worst CTC Grade for Alkaline Phosphatase - All Treated Population
Description: Alkaline Phosphatase was measured as Units per Liter (U/L). National Cancer Institute Common Terminology Criteria (CTC) v3.0 was used to determine Grade. GRADE (1): > 1.0 - 2.5 * upper limits of normal (ULN); GRADE (2): > 2.5 - 5.0 * ULN; GRADE (3): > 5.0 - 20.0 * ULN; GRADE (4): > 20.0 * ULN.
Time Frame: Day 1 to Week 48
Population: Treated participants received at least one dose of a study drug.
Measure: Number; unit: participants
Arm/Group | Paclitaxel, Carboplatin, Ipilimumab | Dacarbazine, Ipilimumab | Ipilimumab
Number analyzed (Participants) | 20 | 19 | 20
participants
  Alkaline Phosphatase Grade 0 | 14 | 18 | 18
  Alkaline Phosphatase Grade 1 | 6 | 1 | 0
  Alkaline Phosphatase Grade 2 | 0 | 0 | 2

26. Secondary Outcome: Number of Participants on Treatment With Toxicity Changes From Baseline by Worst CTC Grade for Total Bilirubin - All Treated Population
Description: Total Bilirubin was measured as milligrams per deciliter (mg/dL). National Cancer Institute Common Terminology Criteria (CTC) v3.0 was used to determine Grade. GRADE (1): > 1.0 - 1.5 * upper limits of normal (ULN); GRADE (2): > 1.5 - 3.0 * ULN; GRADE (3): > 3.0 - 10.0 * ULN; GRADE (4): > 10.0 * ULN.
Time Frame: Day 1 to Week 48
Population: Treated participants received at least one dose of a study drug.
Measure: Number; unit: participants
Arm/Group | Paclitaxel, Carboplatin, Ipilimumab | Dacarbazine, Ipilimumab | Ipilimumab
Number analyzed (Participants) | 20 | 19 | 20
participants
  Total Bilirubin Grade 0 | 20 | 17 | 18
  Total Bilirubin Grade 1 | 0 | 1 | 2
  Total Bilirubin Grade 2 | 0 | 1 | 0

27. Secondary Outcome: Number of Participants on Treatment With Toxicity Changes From Baseline by Worst CTC Grade for Serum Potassium (High) - All Treated Population
Description: Serum potassium was measured as milliequivalents per liter (mEq/L). National Cancer Institute Common Terminology Criteria (CTC) v3.0 was used to determine Grade. GRADE (1): 3.0 - < LLN OR > ULN - 5.5;; GRADE (2): > 5.5 - 6.0; GRADE (3): 2.5 - < 3.0 > 6.0 - 7.0; GRADE (4): < 2.5 mEq/L.
Time Frame: Day 1 to Week 48
Population: Treated participants received at least one dose of a study drug.
Measure: Number; unit: participants
Arm/Group | Paclitaxel, Carboplatin, Ipilimumab | Dacarbazine, Ipilimumab | Ipilimumab
Number analyzed (Participants) | 20 | 19 | 20
participants
  Serum Potassium (High) Grade 0 | 20 | 17 | 17
  Serum Potassium (High) Grade 1 | 0 | 2 | 1
  Serum Potassium (High) Grade 2 | 0 | 0 | 2

28. Secondary Outcome: Number of Participants on Treatment With Toxicity Changes From Baseline by Worst CTC Grade for Total Amylase - All Treated Population
Description: Amylase was measured as units per liter (U/L). National Cancer Institute Common Terminology Criteria (CTC) v3.0 was used to determine Grade. GRADE (1): > 1.0 - 1.5 * upper limits of normal (ULN); GRADE (2): > 1.5 - 2.0 * ULN; GRADE (3): > 2.0 - 5.0 * ULN; GRADE (4): > 5.0 * ULN.
Time Frame: Day 1 to Week 48
Population: Treated participants received at least one dose of a study drug.
Measure: Number; unit: participants
Arm/Group | Paclitaxel, Carboplatin, Ipilimumab | Dacarbazine, Ipilimumab | Ipilimumab
Number analyzed (Participants) | 20 | 19 | 20
participants
  Total Amylase Grade 0 | 20 | 19 | 16
  Total Amylase Grade 1 | 0 | 0 | 2
  Total Amylase Grade 2 | 0 | 0 | 1
  Total Amylase Grade 3 | 0 | 0 | 1

29. Secondary Outcome: Number of Participants on Treatment With Toxicity Changes From Baseline by Worst CTC Grade for Total Calcium (High) - All Treated Population
Description: Total Calcium was measured as milligrams per deciliter (mg/dL). National Cancer Institute Common Terminology Criteria (CTC) v3.0 was used to determine Grade. GRADE (1): 8.0 - < LLN OR > ULN - 11.5; GRADE (2): 7.0 - < 8.0 > 11.5 - 12.5; GRADE (3): 6.0 - < 7.0 > 12.5 - 13.5; GRADE (4): < 6.0 > 13.5 mg/dL.
Time Frame: Day 1 to Week 48
Population: Treated participants received at least one dose of a study drug.
Measure: Number; unit: participants
Arm/Group | Paclitaxel, Carboplatin, Ipilimumab | Dacarbazine, Ipilimumab | Ipilimumab
Number analyzed (Participants) | 20 | 19 | 20
participants
  Total Calcium (High) Grade 0 | 18 | 19 | 19
  Total Calcium (High) Grade 1 | 2 | 0 | 1

30. Secondary Outcome: Number of Participants on Treatment With Toxicity Changes From Baseline by Worst CTC Grade for Total Lipase - All Treated Population
Description: Total Lipase (as measured with a turbidimetric assay) was measured as units per liter (U/L). National Cancer Institute Common Terminology Criteria (CTC) v3.0 was used to determine Grade. GRADE (1): > 1.0 - 1.5 * ULN; GRADE (2): > 1.5 - 2.0 * ULN; GRADE (3): > 2.0 - 5.0 * ULN; GRADE (4): > 5.0 X ULN.
Time Frame: Day 1 to Week 48
Population: Treated participants received at least one dose of a study drug.
Measure: Number; unit: participants
Arm/Group | Paclitaxel, Carboplatin, Ipilimumab | Dacarbazine, Ipilimumab | Ipilimumab
Number analyzed (Participants) | 20 | 19 | 20
participants
  Total Lipase Grade 0 | 12 | 6 | 4
  Total Lipase Grade 1 | 1 | 0 | 0
  Total Lipase Grade 4 | 0 | 0 | 1
  Total Lipase Not Reported | 7 | 13 | 15

31. Secondary Outcome: Number of Participants on Treatment With Toxicity Changes From Baseline by Worst CTC Grade for Uric Acid - All Treated Population
Description: Uric acid was measured as milligrams per deciliter (mg/dL). National Cancer Institute Common Terminology Criteria (CTC) v3.0 was used to determine Grade. GRADE (1): > 1.0 * ULN - 10.0; GRADE (4): > 10.0 mg/dL.
Time Frame: Day 1 to Week 48
Population: Treated participants received at least one dose of a study drug.
Measure: Number; unit: participants
Arm/Group | Paclitaxel, Carboplatin, Ipilimumab | Dacarbazine, Ipilimumab | Ipilimumab
Number analyzed (Participants) | 20 | 19 | 20
participants
  Uric Acid Grade 0 | 20 | 19 | 17
  Uric Acid Grade 1 | 0 | 1 | 3

ADVERSE EVENTS:
Time Frame: Day 1 up to last patient last visit (LPLV) 30 October 2012
Description: Participants continue in the study until disease progression, toxicities requiring discontinuation, withdrawal of consent, or study closure.
Arm/Group | Paclitaxel, Carboplatin, Ipilimumab | Dacarbazine, Ipilimumab | Ipilimumab
Serious Adverse Events (participants affected / at risk) | 12/20 | 10/19 | 14/20
Other Adverse Events (participants affected / at risk) | 20/20 | 19/19 | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Paclitaxel, Carboplatin, Ipilimumab (N=20) | Dacarbazine, Ipilimumab (N=19) | Ipilimumab (N=20)
Asthenia (General disorders) | 1 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hypopituitarism (Endocrine disorders) | 0 | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 | 1 | 2
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 1
Cystitis (Infections and infestations) | 1 | 0 | 0
Fatigue (General disorders) | 2 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 2
Metastases to skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 2 | 1
Meningitis aseptic (Infections and infestations) | 0 | 1 | 0
Radiation necrosis (Injury, poisoning and procedural complications) | 0 | 0 | 1
Autoimmune hepatitis (Hepatobiliary disorders) | 1 | 2 | 0
Autoimmune pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 1
Erythema nodosum (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 0 | 0
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 1
Convulsion (Nervous system disorders) | 0 | 1 | 2
Sepsis (Infections and infestations) | 0 | 0 | 1
Seroma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 2 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 1
Haematemesis (Gastrointestinal disorders) | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Metastases to abdominal cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1
Optic neuritis (Nervous system disorders) | 0 | 0 | 1
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 1
Psychotic disorder (Psychiatric disorders) | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 0 | 1
Bile duct obstruction (Hepatobiliary disorders) | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 1 | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 3 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 4 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Paclitaxel, Carboplatin, Ipilimumab (N=20) | Dacarbazine, Ipilimumab (N=19) | Ipilimumab (N=20)
Autoimmune disorder (Immune system disorders) | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 5 | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0
Generalised oedema (General disorders) | 0 | 0 | 1
Gingival inflammation (Gastrointestinal disorders) | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1 | 0
Haemoglobin decreased (Investigations) | 11 | 7 | 4
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 2 | 0 | 1
Hypopituitarism (Endocrine disorders) | 1 | 0 | 1
Incision site complication (Injury, poisoning and procedural complications) | 0 | 0 | 1
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Migraine (Nervous system disorders) | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0
Neurodermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Oesophageal pain (Gastrointestinal disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Procedural headache (Injury, poisoning and procedural complications) | 0 | 1 | 0
Rocky mountain spotted fever (Infections and infestations) | 0 | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 2
Abdominal hernia (Gastrointestinal disorders) | 1 | 0 | 0
Amylase increased (Investigations) | 2 | 2 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 2
Aspartate aminotransferase increased (Investigations) | 5 | 10 | 3
Bacterial infection (Infections and infestations) | 0 | 0 | 1
Blood albumin decreased (Investigations) | 1 | 0 | 1
Chest pain (General disorders) | 1 | 0 | 0
Chromaturia (Renal and urinary disorders) | 0 | 1 | 0
Discomfort (General disorders) | 0 | 0 | 1
Fatigue (General disorders) | 12 | 18 | 12
Flatulence (Gastrointestinal disorders) | 2 | 2 | 1
Generalised erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 2 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 7 | 2 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Infection (Infections and infestations) | 0 | 1 | 0
Malaise (General disorders) | 0 | 2 | 0
Oral pain (Gastrointestinal disorders) | 0 | 1 | 0
Radial nerve palsy (Nervous system disorders) | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Spinal pain (General disorders) | 0 | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 1
Tooth infection (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 1 | 2
Vision blurred (Eye disorders) | 2 | 1 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 3 | 3
Agitation (Psychiatric disorders) | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 12 | 1 | 3
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 6 | 2
Bladder pain (Renal and urinary disorders) | 0 | 0 | 1
Blood corticotrophin decreased (Investigations) | 0 | 0 | 1
Blood testosterone decreased (Investigations) | 0 | 1 | 1
Body tinea (Infections and infestations) | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 2 | 2
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1
Libido decreased (Psychiatric disorders) | 0 | 1 | 1
Mass (General disorders) | 0 | 1 | 0
Movement disorder (Nervous system disorders) | 0 | 0 | 1
Mucosal inflammation (General disorders) | 2 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 4 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 5
Ocular discomfort (Eye disorders) | 0 | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 1 | 0 | 1
Panic attack (Psychiatric disorders) | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 0
Photophobia (Eye disorders) | 0 | 1 | 0
Platelet count decreased (Investigations) | 10 | 5 | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Renal pain (Renal and urinary disorders) | 0 | 1 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Sinus headache (Nervous system disorders) | 0 | 1 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0 | 1
Visual impairment (Eye disorders) | 0 | 1 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 0 | 1
Autoimmune hepatitis (Hepatobiliary disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 4 | 3
Blood creatinine increased (Investigations) | 1 | 2 | 2
Blood phosphorus decreased (Investigations) | 0 | 0 | 1
Candidiasis (Infections and infestations) | 0 | 0 | 2
Chills (General disorders) | 3 | 3 | 2
Cyanosis (Cardiac disorders) | 1 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 2
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Eye pain (Eye disorders) | 1 | 0 | 0
Faecal incontinence (Gastrointestinal disorders) | 0 | 0 | 1
Flat affect (Psychiatric disorders) | 0 | 0 | 1
Folliculitis (Infections and infestations) | 1 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 1
Insomnia (Psychiatric disorders) | 3 | 6 | 7
Menstruation irregular (Reproductive system and breast disorders) | 0 | 1 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Mydriasis (Eye disorders) | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1
Nodule (General disorders) | 1 | 0 | 0
Olfactory nerve disorder (Nervous system disorders) | 1 | 0 | 0
Pain (General disorders) | 3 | 1 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 3 | 2
Scar (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 1 | 0
Tinea cruris (Infections and infestations) | 0 | 0 | 1
Tinea pedis (Infections and infestations) | 1 | 0 | 1
Uveitis (Eye disorders) | 1 | 1 | 0
Waist circumference increased (Investigations) | 0 | 0 | 1
Weight increased (Investigations) | 1 | 0 | 1
White blood cell count decreased (Investigations) | 10 | 2 | 1
Anxiety (Psychiatric disorders) | 1 | 2 | 2
Ataxia (Nervous system disorders) | 0 | 0 | 1
Convulsion (Nervous system disorders) | 0 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 0
Dry eye (Eye disorders) | 0 | 1 | 1
Early satiety (General disorders) | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 2 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 5 | 0 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 1 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 1
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 2 | 0
Neutrophil count decreased (Investigations) | 10 | 4 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Onychomycosis (Infections and infestations) | 0 | 1 | 0
Oral herpes (Infections and infestations) | 0 | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Salmonellosis (Infections and infestations) | 0 | 1 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Sleep disorder (Psychiatric disorders) | 1 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Vitiligo (Skin and subcutaneous tissue disorders) | 2 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 4 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0
Blood cortisol decreased (Investigations) | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 10 | 12 | 12
Diplopia (Eye disorders) | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 4 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 2 | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Gait disturbance (General disorders) | 0 | 0 | 1
Gout (Metabolism and nutrition disorders) | 0 | 0 | 2
Headache (Nervous system disorders) | 7 | 10 | 6
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 2 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 10 | 4 | 5
Infusion site pain (General disorders) | 0 | 1 | 0
Lentigo maligna (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 1 | 0
Mucous membrane disorder (General disorders) | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2
Nausea (Gastrointestinal disorders) | 12 | 15 | 7
Oedema peripheral (General disorders) | 4 | 2 | 3
Papule (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Periorbital oedema (Eye disorders) | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Sinusitis (Infections and infestations) | 0 | 2 | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 6 | 3
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Angiosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Bartholin's cyst (Reproductive system and breast disorders) | 0 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 6 | 5 | 1
Cataract (Eye disorders) | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 1
Constipation (Gastrointestinal disorders) | 8 | 10 | 7
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 2
Dysgeusia (Nervous system disorders) | 4 | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 12 | 6 | 5
Hypersensitivity (Immune system disorders) | 6 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 5 | 2 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypophysitis (Endocrine disorders) | 0 | 2 | 5
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Lymphoedema (Vascular disorders) | 0 | 0 | 1
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Oedema (General disorders) | 0 | 1 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 0 | 0
Photopsia (Eye disorders) | 0 | 1 | 1
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 1 | 0
Pyrexia (General disorders) | 5 | 8 | 4
Rash (Skin and subcutaneous tissue disorders) | 16 | 11 | 17
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 2 | 2
Weight decreased (Investigations) | 2 | 4 | 3
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Wound complication (Injury, poisoning and procedural complications) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 5 | 7 | 4
Adrenal insufficiency (Endocrine disorders) | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 5 | 10 | 3
Auricular perichondritis (Ear and labyrinth disorders) | 0 | 0 | 1
Blood uric acid increased (Investigations) | 0 | 0 | 1
Catheter site discharge (General disorders) | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 0 | 2
Decreased appetite (Metabolism and nutrition disorders) | 6 | 8 | 5
Depression (Psychiatric disorders) | 1 | 3 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 2 | 0
Eye inflammation (Eye disorders) | 0 | 0 | 1
Flushing (Vascular disorders) | 3 | 5 | 1
Hemiparesis (Nervous system disorders) | 0 | 0 | 1
Hyperalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 1 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0 | 0
Lipase increased (Investigations) | 3 | 4 | 1
Mechanical urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 9 | 1 | 2
Occult blood positive (Investigations) | 0 | 1 | 0
Odynophagia (Gastrointestinal disorders) | 1 | 0 | 0
Oxygen saturation decreased (Investigations) | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 13 | 14 | 15
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 1
Temperature intolerance (General disorders) | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 2 | 1
Tooth abscess (Infections and infestations) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 5 | 8 | 6
Xerosis (General disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.